CLINICAL TRIAL: NCT02266095
Title: Pilot Study of a Novel Splint Treatment for Thumb CMC Joint Arthritis: a Comparison of Oval-8 Splinting Versus Standardized Treatment With Tee Pee or Forearm Based Thumb Spica Splinting
Brief Title: Oval-8 Splinting Versus Standardized Treatment With Tee Pee or Forearm Based Thumb Spica Splinting
Acronym: Oval-8
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed prior to enrolling patients
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UFJ 2013-136
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2015-12

CONDITIONS: Carpometacarpal (CMC) Joint Arthritis
Keywords: Osteoarthritis; Thumb spica splint; Oval-8 splint; Tee-Pee splint
MeSH Terms: conditions — Capillary Malformations, Congenital, 1; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oval-8 Splint (Active Comparator): Patients will be asked to wear their assigned splint 24 hours per day with removal for hygiene care. Follow-up appointments will occur at week 4 and 12. Each visit will include a clinical examination, splint assessment for continued appropriate fit and evaluation of skin for irritation or breakdown.
  Standard non-operative therapy includes activity modification, therapy, NSAIDS, splinting (thumb spica or Tee-Pee). Oval-8 splints are not commonly used for treatment of thumb CMC arthritis.
  Procedures will be undertaken to minimize patient discomfort. Participants will be instructed to continue with range of motion exercises to 2-5th digits and elbow to try to avoid stiffness.
  Interventions: Device: Oval-8 Splint
- Tee Pee Splint (Active Comparator): Patients will be asked to wear their assigned splint 24 hours per day with removal for hygiene care. Follow-up appointments will occur at week 4 and 12. Each visit will include a clinical examination, splint assessment for continued appropriate fit and evaluation of skin for irritation or breakdown.
  Standard non-operative therapy includes activity modification, therapy, NSAIDS, splinting (thumb spica or Tee-Pee).
  Procedures will be undertaken to minimize patient discomfort. Participants will be instructed to continue with range of motion exercises to 2-5th digits and elbow to try to avoid stiffness.
  Interventions: Device: Tee Pee Splint
- Forearm Based Splint (Active Comparator): Patients will be asked to wear their assigned splint 24 hours per day with removal for hygiene care. Follow-up appointments will occur at week 4 and 12. Each visit will include a clinical examination, splint assessment for continued appropriate fit and evaluation of skin for irritation or breakdown.
  Standard non-operative therapy includes activity modification, therapy, NSAIDS, splinting (thumb spica or Tee-Pee).
  Procedures will be undertaken to minimize patient discomfort. Participants will be instructed to continue with range of motion exercises to 2-5th digits and elbow to try to avoid stiffness.
  Interventions: Device: Forearm Based Splint

INTERVENTIONS:
Device: Oval-8 Splint — Splinting with Oval-8
  Arms: Oval-8 Splint
Device: Tee Pee Splint — Splinting with Tee Pee
  Arms: Tee Pee Splint
Device: Forearm Based Splint — Splinting with Forearm based
  Arms: Forearm Based Splint

SUMMARY:
The oval-8 splint has been developed for many uses in finger pathology and trauma. It has not, however, been used to treat thumb carpometacarpal (CMC) joint arthritis. When treating thumb CMC joint osteoarthritis, splinting is a very widely used and supported treatment option for non-operative management. Many studies have been performed showing that thumb spica splinting in abduction with either a hand based or forearm based splint improves pain. This study aims to compare the effects of a novel splinting approach with oval-8 splints for the hyperextended thumb interphalangeal (IP) joint vs. standardized treatment with Tee Pee splinting (hand based thumb spica) or forearm thumb spica splinting on pain and function of patients with thumb CMC joint arthritis.

This is a pilot study will address the following hypothesis: Splinting of the hyperextended thumb IP joint with oval-8 splints will lead to increased DASH scores and decreased pain on physical exam compared to splinting with thumb spica splints in patients with thumb CMC arthritis.

DETAILED DESCRIPTION:
After informed consent is obtained and the patient has met all of the inclusion criteria and non of the exclusion criteria, the patient will be assigned a study ID number. The patient will be randomized with a ratio of 1:1:1 to a splint treatment with either a forearm thumb spica splint, Tee-Pee splint or oval- 8 splint at the time of initial visit to Orthopaedic Hand clinic (week 1 visit). The patient will be fitted and provided with the appropriate splint by Orthopaedic physician.

Baseline radiographs (3 views anterior-posterior, lateral and oblique) and data points will be gathered from initial clinic history and physical, as performed per normal clinical protocol: arthritis grade, hand involved, dominant hand, interphalangeal (IP) extension, MCP extension, pinch strength, grip strength, pain scale, location of pain, DASH scores, analgesic use, and work/hobby activity. Additionally, demographic data including age, gender and race/ethnicity will be gathered and patient will be asked to repeat pinch and grip tests with study splint applied and asked to repeat assessment of pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Carpometacarpal (CMC) osteoarthritis
* greater than or equal to 35 degrees of passive thumb interphalangeal (IP) joint hyperextension on physical exam

Exclusion Criteria:

* History of hand surgery to affected hand
* Prior surgical treatment for thumb carpometacarpal (CMC) osteoarthritis.
* Patients with diagnosis of an autoimmune arthritis and post traumatic arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
DASH Score | 12 Weeks
  The DASH is scored in two components. The disability/symptom questions (30 items scored 1-5) includes the following scoring categories: no difficulty - unable, not at all - extremely, not limited at all - unable, none - extreme, no difficulty - so much difficulty that I can't sleep, and strongly disagree - strongly agree. At least 27 out of 30 items must be completed for a score to be calculated. The assigned values for all completed responses are summed and averaged, producing a score out of five.
  The second section high performance sport/music or work section. This section of 4 items scored 1-5 includes no difficulty - unable, scoring category. The scoring calculations are the same for this area.

SECONDARY OUTCOMES:
Pain Score | 12 Weeks
  The general pain scale ranges 0 - 10, with 0 being no pain and 10 being worst possible pain. Pinch pain and Grip pain will the measured with and without the splint. The ranges are the same for all pain scales.

CONTACTS AND LOCATIONS:
Overall Officials: Marc B Kaye, M.D., Principal Investigator — University of Florida
Locations (1):
- UF Health Orthopaedics - Jacksonville (Emerson), Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share participant data as no patients were enrolled in the study.